CLINICAL TRIAL: NCT01384903
Title: An Open-label Study of KW-3357 Compared to Plasma-derived Antithrombin for Disseminated Intravascular Coagulation (DIC) Associated With Infection
Brief Title: An Open-label Study of KW-3357
Acronym: 3357-004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3357-004
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Disseminated Intravascular Coagulation (DIC)
MeSH Terms: conditions — Disseminated Intravascular Coagulation

ARMS (2):
- KW-3357 (Experimental)
  Interventions: Drug: KW-3357
- Plasma-derived antithrombin (Active Comparator)
  Interventions: Drug: Plasma-derived antithrombin

INTERVENTIONS:
Drug: KW-3357 — Intravenous infusion once a day
  Arms: KW-3357
Drug: Plasma-derived antithrombin — Intravenous infusion once a day
  Arms: Plasma-derived antithrombin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KW-3357 compared to plasma-derived antithrombin using multi-center, open-label, parallel-group, comparative method in patients with Disseminated Intravascular Coagulation (DIC) associated with infection.

ELIGIBILITY:
Inclusion Criteria:

* Meet the ACCP/SCCM-defined sepsis criteria
* Japanese Association for Acute Medicine-defined DIC criteria score >= 4
* Antithrombin activity <= 70%
* Written informed consent from patient or guardian

Exclusion Criteria:

* Anamnesis or complication of serious drug allergy
* Serious liver disorder, such as fulminant hepatitis and decompensated cirrhosis
* Pregnant, nursing, or possibly pregnant woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
DIC resolution | 6 days (or discontinuation)
  Japanese Association for Acute Medicine-defined DIC criteria score < 4

SECONDARY OUTCOMES:
DIC score | Screening, 2, 3, 4, 5, 6 days (or discontinuation)
  Based on the Japanese Association for Acute Medicine-defined DIC criteria score
Mortality | 28 days
Organ symptoms | Screening, 4, 6 days (or discontinuation)
  Sepsis related organ failure assessment score
Severity | Screening, 4, 6 days (or discontinuation)
  The Acute Physiology and Chronic Health Evaluation II score
Plasma antithrombin activity | Screening, 2, 3, 4, 5, 6 days (or discontinuation)
Number of patients with adverse events | up to 6 days (or discontinuation)

CONTACTS AND LOCATIONS:
Locations (1):
- Saga, Japan

REFERENCES:
- [Derived] Endo S, Shimazaki R; Antithrombin Gamma Study Group. An open-label, randomized, phase 3 study of the efficacy and safety of antithrombin gamma in patients with sepsis-induced disseminated intravascular coagulation syndrome. J Intensive Care. 2018 Nov 16;6:75. doi: 10.1186/s40560-018-0339-z. eCollection 2018. PMID 30473794